CLINICAL TRIAL: NCT07301424
Title: Phase II Study of Subcutaneous Blinatumomab Plus Ponatinib for BCR-ABL Positive B-Cell Acute Lymphoblastic Leukemia
Brief Title: Subcutaneous Blinatumomab Plus Ponatinib for BCR-ABL+ B-ALL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLSG-ALL-2
Record Dates: First submitted 2025-12-12; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia (ALL) Philadelphia Chromosome-positive (Ph+); BCR-ABL Positive Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; Ponatinib; BiTE antibody; Acute lymphoblastic leukemia; BCR-ABL positive acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with subcutaneous blinatumomab plus ponatinib (Experimental)
  Interventions: Drug: Treatment with blinatumomab given subcutaneously.

INTERVENTIONS:
Drug: Treatment with blinatumomab given subcutaneously. — Previous studies have used intravenous blinatumomab combined with a TKI (ponatinib or dasatinib) for patients with BCR-ABL positive B-ALL. This study is using subcutaneous blinatumomab combined with ponatinib for previously untreated patients with this disease.

SUMMARY:
B-cell acute lymphoblastic leukemia (B-ALL) is an aggressive blood cancer; about 30% of B-ALL cases in adults have a mutation called BCR-ABL that drives the disease.

Blinatumomab is an antibody drug that targets B-ALL cells and helps the immune system to kill them. It is usually given intravenously, but a newer formulation can be given under the skin. Ponatinib is a drug, taken by mouth, that targets and kills leukemia cells that have the BCR-ABL mutation.

The goal of this clinical trial is to test the effectiveness of treating patients with BCR-ABL positive B-ALL with blinatumomab given subcutaneously (under the skin) combined with ponatinib tablets. The study will also evaluate what side effects occur using this combination.

Participants will first receive ponatinib tablets for 70 days, along with prednisone for the first month. This will be followed by blinatumomab injections 3 times per week for 4 weeks, repeated for 5 treatment cycles, along with ponatinib. Participants will then continue ponatinib tablets alone for 5 years from the start of treatment.

During treatment, participants will undergo regular blood and bone marrow tests to see how well the treatment is working, and to check for side effects. The effect of this treatments on their quality of life will also be evaluated.

DETAILED DESCRIPTION:
This Phase II clinical trial will evaluate with efficacy and tolerance of subcutaneous (sc) blinatumomab (blina) combined with ponatinib for previously untreated patients with BCR-ABL (Ph) positive B-cell acute lymphoblastic leukemia (ALL).

Participants will, after a brief steroid pre-phase, receive induction therapy with ponatinib 30 mg/day x 70 days, with prednisone for the first month. They will then receive 5 cycles of consolidation therapy with sc blina. The first cycle will consist of blina 250 mcg sc daily x 7 days, then 500 mcg sc 3x/week x 3 weeks. Cycles 2-5 will consist of blina 500 mcg sc 3x/week x 4 weeks. There will be a 2 week break in between each consolidation cycle. Ponatinib will continue at 30 mg daily through the end of consolidation. Participants will then receive maintenance therapy with ponatinib 15 mg/day until 5 years from the start of induction.

Intrathecal chemotherapy will be administered for a total of 15 doses; this will include 7 doses during induction, 1 dose in between each consolidation cycle, and 4 during maintenance.

Efficacy will be determined by bone marrow assessments for MRD at various timepoints. The primary endpoint is the measurable residual disease (MRD) response after the end of consolidation cycle 2, by both BCR-ABL PCR (MRD4 or greater) and by IgR (MRD negativity by Clonoseq[R]). The CR rate, MRD response duration, RFS and OS will also be assessed.

Toxicity will be evaluated throughout the study and graded using CTCAE V5. Quality of life will be assessed at various timepoints using QLQ-C30.

ELIGIBILITY:
Inclusion Criteria:

1. Ph positive [either t(9;22) and/or BCR-ABL1 positive] ALL, CD19 positive
2. Age ≥18 years at time of informed consent
3. No prior induction treatment for ALL. A brief corticosteroid pre-phase (< 1 week), or hydroxyurea for cytoreduction or symptom control is permitted.

3. Greater than or equal to 5% blasts in the BM.

4. Performance status ≤2 (ECOG Scale, see Appendix IV)

5. Adequate organ function: 5.1.5.1 Hepatic:

Adequate liver function as defined by the following criteria (unless the increased values are judged to be leukemia disease related):

Total serum bilirubin less than 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome or Meulengracht disease Alanine aminotransferase (ALT) less than 3 x ULN Aspartate aminotransferase (AST) less than 3 x ULN 5.1.5.2 Pancreatic:

* Serum lipase less than 2 x ULN 5.1.5.3 Renal:
* Estimated Creatinine clearance ≥ 40 mL/min 5.1.5.4 Cardiac:
* Left ventricular ejection fraction > 40%

Exclusion Criteria:

1. Uncontrolled infection
2. Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus
3. Presence of cardiovascular disease of clinical relevance within the past 3 months. This includes:

   5.2.3.1 Unstable angina 5.2.3.2 Myocardial infarction 5.2.3.3 Transient ischemic attack or stroke 5.2.3.4 Peripheral vascular infarction, claudication and/or revascularization 5.2.3.5 Symptomatic congestive heart failure 5.2.3.6 Clinically significant significant atrial/ventricular tachyarrhythmias 5.2.3.7 Venous thromboembolic event requiring systemic anticoagulation

   Please consult the sponsor if there are specific concerns outside of these criteria
4. Uncontrolled hypertension
5. History or presence of clinically relevant CNS pathology or event.

   This may include, for example:

   epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome or psychosis.

   Before excluding a potential subject, please consult the sponsor.
6. Any other concurrent disease or medical condition that could be exacerbated by the treatment or would seriously complicate compliance with the protocol.
7. History of malignancy other than ALL within 3 years prior to start of protocol-specified therapy except for:

   * malignancy treated with curative intent and with no known active disease present for 3 years before enrollment, and felt to be at low risk for recurrence by the treating physician
   * adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * adequately treated cervical carcinoma in situ without evidence of disease
   * adequately treated breast ductal carcinoma in situ without evidence of disease
   * prostatic intraepithelial neoplasia without evidence of prostate cancer
8. Prior hematologic malignancy and/or alloSCT; this includes known CML
9. Concurrent or prior (within 30 days) treatment with another investigational agent or study drug
10. Female subject is pregnant or breastfeeding or planning to become pregnant breastfeed during treatment, and for an additional 4 months after the last dose of protocol-specified therapy
11. Inability to swallow or absorb tablets
12. Subject considered unsuitable for study for any other reason in the physician's best judgement. Before excluding a potential subject, please consult the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
• MR4 rate for BCR-ABL1 by PCR after 2 cycles of blinatumomab | At end of cycle 2 of blinatumomab (each cycle is 28 days).
  After 2 cycles of blinatumomab, the bone marrow will be tested for MRD by PCR for BCR-ABL. The rate of MRD4 (MRD<10[-4]) at this timepoint will constitute a primary outcome.
Complete molecular response (CMR) by IgR (Clonoseq[R]) after 2 cycles of blinatumomab. | At end of cycle 2 of Blinatumomab (each cycle being 28 days).
  After 2 cycles of Blinatumomab the marrow will be tested for MRD by Clonoseq. The rate of MRD negativity by IgR will constitute a primary outcome.

SECONDARY OUTCOMES:
Complete response rate | Determined at the end of the 70 day induction phase
  Complete response rate (CR and CRh) of ponatinib + prednisone
Patient and caregiver experience | At screening, end of induction (Day 70), end of cycles 2 and 5 of blinatumomab, and one year after start of maintenance therapy with ponatinib.
  EORTC QLQ-C30 scores
Molecular response duration | From the time of documented remission at Day 70 of induction, until the date of first documented molecular progression, assessed up to 5 years from the start of treatment.
  The duration of MR4 by PCR and CMR by Clonoseq will be determined in follow-up bone marrow assessments.
Relapse-free survival (RFS) | From the date of documented remission at day 70 until the date of first documented relapse or date of death from any cause, whichever came first, assessed up to 5 years from the start of treatment.
  Time from primary outcome to molecular disease progression.
Overall survival (OS) | From the date of enrollment until the date of death from any cause or last follow-up, assessed up to 5 years from the start of treatment.
  Time from start of treatment until death form any cause or last follow-up.
Safety and tolerability | From the start of study treatment through the completion of study treatment at 5 years.
  Safety and tolerability of the ponatinib plus blinatumomab combination, based on TEAE's, graded by CTCAE V5, as well as by CRS and ICANS grading.
Prognostic factors for remission | At the primary endpoint at the end of cycle 2 of blinatumomab (each cycle being 28 days).
  Correlation of primary efficacy endpoints (MR4, CMR) with diagnostic NGS, IKZFplus genotype, age and baseline WBC
Prognostic factors for relapse-free survival | From date of documented remission at day 70 of induction, until the date of relapse or date of death from any cause, whichever came first, assessed up to 5 years.
  Correlation of RFS with diagnostic NGS, IKZFplus genotype, age and baseline WBC
Prognostic factors for overall survival | From date of enrollment until the date of death from any cause or last follow-up, assessed up to 5 years.
  Correlation of OS with diagnostic NGS, IKZFplus genotype, age and baseline WBC

OTHER OUTCOMES:
Exploratory: comparison of different MRD outcomes | After the completion of cycle 2 of blinatumomab (each cycle being 28 days).
  Concordance between MRD results in bone marrow by BCR-ABL PCR vs IgR vs flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) regarding baseline molecular data and molecular response data collected in this study will be made available to other researchers on request.
Time Frame: These data will be made available once the primary outcome data on all subjects are available, and after results have been reported and published.
Access Criteria: Academic researchers may be provided with the data on request only.